CLINICAL TRIAL: NCT02375919
Title: The Pulmonary Embolism Rule Out Criteria (PERC) Rule to Exclude the Diagnosis of Pulmonary Embolism in Emergency Low Risk Patients: a Non-inferiority Randomized Controlled Trial
Brief Title: PERC Rule to Exclude Pulmonary Embolism in the Emergency Deparment
Acronym: PROPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IDRCB 2015-A00215-44; P1409 (Other: AP-HP)
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Emergency Patients
Keywords: PERC rule; emergency department; pulmonary embolism
MeSH Terms: conditions — Emergencies; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Emergency physician will assess low risk patients for PE with conventional strategy, using D-Dimer testing with subsequent CTPA if positive
- Intervention (Other): PERC based Strategy : Emergency physician will assess low risk patients for PE first with calculation of PERC score. If all PERC criteria are negative, then no further testing for PE is recommended. If at least one criterion is positive, then the patient undergoes D-Dimer testing with subsequent CTPA if positive
  Interventions: Other: PERC based Strategy

INTERVENTIONS:
Other: PERC based Strategy — work up for diagnosis of PE includes calculation of PERC
  Arms: Intervention

SUMMARY:
The Pulmonary Embolism Rule Out Criteria (PERC) is an 8-item rule, that was derived and tested to rule out the diagnosis of Pulmonary Embolism (PE) in the Emergency Department (ED) amongst low risk patients. Even though meta analyses have confirmed the safety of its utilization, equipoise remains - especially in European country where the prevalence of PE is higher than in the US- on whether this rule could be safely applied to all low risk emergency patients with a suspicion of PE.

The PROPER Trial is a non inferiority , cluster randomized trial. All centers will recruit patients with a suspicion of PE and a low pre test probability. To rule out the diagnosis of PE, center will use the usual diagnostic strategies with D-dimeres measurement for 6 months, and PERC based strategy for 6 months.

In the control group (usual strategy), patients will be tested for D-dimeres, followed if positive by a Computed Tomography of Pulmonary Artery (CTPA).

In the intervention group (PERC Based), patients will be first assessed with PERC score. If PERC=0, then the diagnosis of PE will be exclude with no supplemental investigations. If PERC>0, then patients will undergo the usual strategy, with D-dimeres measurement +/- CTPA.

The primary outcome is the failure percentage of the diagnostic strategy, defined as diagnosed deep venous thrombosis (DVT) or PE at 3 month follow up, among patients for whom PE has been initially ruled out.

DETAILED DESCRIPTION:
The diagnosis of Pulmonary Embolism (PE) in the Emergency Department (ED) is crucial. As emergency physicians fear to miss this potential lethal condition, PE tends to be overdiagnosed with potential source of unnecessary risks and no clear benefit in terms of outcome. PERC is an 8-item block of clinical criteria that can identify patients who can safely be discharged without further investigation in the ED for the diagnosis of PE. The endorsement of this rule could markedly reduce the number of irradiative imaging studies, length of stay in the ED, and rate of adverse event resulting from both diagnostic and therapeutic means. Several retrospective and prospective studies have shown the safety and benefits of PERC rule for PE diagnosis in low risk patients. However, no randomized study has yet compared the benefit/risk ratio of PERC based strategy with the standard diagnosis strategy and thus validated its endorsement in this setting. We hypothesize that in patients with a low gestalt clinical probability and a PERC negative, PE can be safely ruled out and the patient discharged with no further testing

This is a controlled, cluster randomized trial in Europe (N=15). Each center will be randomized on the sequence of period intervention: 6 months intervention (PERC based strategy) followed by 6 months control (usual care), or 6 months control followed by 6 months intervention with 2 months of "wash-out" between the two periods.

The primary objective of this study is to assess the non inferiority of a PERC based diagnosis strategy for PE low risk emergency patients, compared to the standard strategy of D-dimer testing, on the occurrence of non-diagnosed thrombo-embolic event.

The primary outcome is the failure percentage of the diagnostic strategy, defined as diagnosed DVT or PE at 3 month follow up, among patients for whom PE has been initially ruled out. Exclusion of PE in the ED is made upon negative D-dimere result or negative CTPA in both groups, or negative PERC in the intervention group.

Secondary objectives are :

To assess the reduction of unnecessary irradiative imaging studies and adverse events. To assess the reduction in ED length of stay, undue onset of anticoagulation regimen and associated adverse events. To assess the reduction of hospital admission, readmission, and mortality at 3 months.

Secondary endpoints include:

* Rate of CTPA and related adverse events
* Length of stay in the ED (hours)
* Anticoagulant therapy administration and adverse events
* Admission to the hospital following ED visit.
* All causes re hospitalization at 3 months,
* Death from all causes at 3 months

The two groups will have a different work up for the diagnosis of PE in the ED as follows:

Experimental group:

PERC based strategy: work up for diagnosis of PE includes calculation of PERC. If all PERC criteria are negative, no further testing for PE is recommended. If at least one criterion is positive, then the patient undergoes sensitive D-dimer testing, with subsequent CTPA if positive. In case of negative D-dimer result, PE will be excluded.

Control group:

Standard strategy: conventional work up for diagnosis of PE. Every low risk patient will undergo sensitive D-dimer testing, with subsequent CTPA if positive. In case of negative D-dimer, PE will be excluded.

All patients with chest pain or dyspnea will be screened and included in the ED by emergency physicians and research assistant. If the treating emergency physician or local investigator considers that the patient has a sufficient clinical suspicion of PE that he needs formal work up for this diagnosis, and that this suspicion is low enough to discard this suspicion in case of negative D-dimer, then the patient will be eligble and asked for written informed consent.

When recruiting a patient, the emergency physician or local investigator will have to confirm in written that he answered "yes" to the two following sentences:

This patient has a clinical suspicion of Pulmonary Embolism, and this diagnosis needs to be formally ruled out or confirmed before discharge I estimate the empirical clinical probability of Pulmonary Embolism as low

After written informed consent has been obtained, the patient can be included in the study.

Included patients will be followed up by phone interview or hospital visit at three months (13 weeks) by a clinical research technician. The time frame of three months could be subject to minor adjustement, and will occur between day 84 and day 98. Follow up visit or interview will seek the occurrence of thrombo-embolic event (DVT documented with ultrasonography of the lower limbs or venous CT, or PE documented with positive CTPA or high probability V/Q lung scan), death, return visit to the ED, hospitalisation.

All medical record pertaining to the patient from this timeframe will be sought and analysed by the local investigator, to found report of thrombo-embolic event, or adverse events from CTPA or anticaogulation. In the cases of death, or report of a thrombo-embolic event, the file will be analysed by a comitee of three independent experts.

This method of adjudication has been described and validated in all major previous diagnostic studies on PE.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of, or worsening of dyspnea Or chest pain
* Low clinical pretest probability of PE, empiricially estimated by the gestalt.

Exclusion Criteria:

* Other obvious cause than PE for dyspnea or chest pain
* Acute severe presentation
* Contra-indication to CTPA
* Concurrent anticoagulation treatment
* Current diagnosed thrombo-embolic event
* Inability to follow up
* Prisoners
* Pregnancy
* No social security
* Participation in another intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1922 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Failure percentage of the diagnostic strategy (diagnosed deep venous thrombosis or pulmonary embolism) at 3 month follow up | 3 months

SECONDARY OUTCOMES:
Rate of Computed Tomography Pulmonary Angiogram (CTPA) and related adverse event | 3 months
  Rate of CTPA related adverse events, defined as anaphylactoid reaction requiring therapeutic intervention within 24 hours, and contrast induced nephropathy with documented >25% increase in creatinine level within three months
Length of stay in the Emergency Department | From date of entry in the emergency department to date of exit
Anticoagulation therapy administration (number of day with treatment within three months) | 3 months
Rate of patients admitted in the hospital following Emergency Department visit | 3 months
All causes re hospitalization at 3 months | 3 months
Death from all causes at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan Freund, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Freund Y, Cachanado M, Aubry A, Orsini C, Raynal PA, Feral-Pierssens AL, Charpentier S, Dumas F, Baarir N, Truchot J, Desmettre T, Tazarourte K, Beaune S, Leleu A, Khellaf M, Wargon M, Bloom B, Rousseau A, Simon T, Riou B; PROPER Investigator Group. Effect of the Pulmonary Embolism Rule-Out Criteria on Subsequent Thromboembolic Events Among Low-Risk Emergency Department Patients: The PROPER Randomized Clinical Trial. JAMA. 2018 Feb 13;319(6):559-566. doi: 10.1001/jama.2017.21904. PMID 29450523
- [Derived] Freund Y, Rousseau A, Guyot-Rousseau F, Claessens YE, Hugli O, Sanchez O, Simon T, Riou B. PERC rule to exclude the diagnosis of pulmonary embolism in emergency low-risk patients: study protocol for the PROPER randomized controlled study. Trials. 2015 Nov 25;16:537. doi: 10.1186/s13063-015-1049-7. PMID 26607669